CLINICAL TRIAL: NCT06087094
Title: Randomized, Double-blind, Placebo-controlled, Single-dose Ascending Study for the Assessment of Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of HRS-7450 in Healthy Subjects.
Brief Title: A Trial of HRS-7450 in Chinese Healthy Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fujian Shengdi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HRS-7450-101
Record Dates: First submitted 2023-10-09; First posted 2023-10-17 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Cerebral Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Cohor 1: HRS-7450 dose 1 or Placebo; (Experimental)
  Interventions: Drug: HRS-7450 ；Placebo
- Cohor 1: HRS-7450 dose 2 or Placebo; (Experimental)
  Interventions: Drug: HRS-7450 ；Placebo
- Cohor 1: HRS-7450 dose 3 or Placebo; (Experimental)
  Interventions: Drug: HRS-7450 ；Placebo
- Cohor 1: HRS-7450 dose 4 or Placebo; (Experimental)
  Interventions: Drug: HRS-7450 ；Placebo
- Cohor 1: HRS-7450 dose 5 or Placebo; (Experimental)
  Interventions: Drug: HRS-7450 ；Placebo

INTERVENTIONS:
Drug: HRS-7450 ；Placebo — HRS-7450 or Placebo

SUMMARY:
The purpose of this First-in-Human study is to evaluate the safety and tolerability after single ascending doses of HRS-7450 given to healthy subjects, compared to placebo..

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female subjects between 18 and 45 years of age (inclusive) at the screening visit
2. Female weighed ≥ 45 kg, male weighed ≥ 50 kg, and all weighed ≤ was 90 kg, and a BMI between 18-28 kg/m²(inclusive)
3. Subjects with fertility promised to have no fertility, sperm or egg donation plan and voluntarily take efficient contraceptive measures ( including partners ) within two weeks before screening and 6 months after the last administration
4. Able to provide written, informed consent prior to initiation of any trial-related procedures, and able, in the opinion of the Principal Investigator, to comply with all the requirements of the trial

Exclusion Criteria:

1. Subjects with a history of drug allergy, or a history of allergy ( asthma, urticaria, eczema, etc. ), or allergic constitution ( such as allergies to two or more drugs, food, and pollen ) or intolerance to any ingredients of the study drug
2. Subjects with heart, respiration, endocrine, metabolism, kidney, liver, gastrointestinal tract, skin, infection, malignant tumor, blood, nervous system disease or mental illness, metabolic dysfunction prior to screening or administration
3. The results of physical examination, vital sign examination, laboratory examination, etc. during the screening are deemed clinically significant
4. Subjects with risk factors for torsades de pointes ventricular tachycardia, or had a family history of short QT syndrome, long QT syndrome, unexplained sudden death in youth ( ≤ 40 years old ), drowning or sudden infant death syndrome in first-degree relatives ( i.e., biological parents, siblings or children )
5. Subjects with hyperkalemia, hypokalemia, hypermagnesemia, hypomagnesemia, hypercalcemia or hypocalcemia are deemed clinically significant
6. ECG examination is clinical significant, such as QTcF > 470ms
7. Subjects with gastrointestinal, urinary and other bleeding tendencies or other high-risk bleeding tendencies within 3 weeks before screening; or those who have arterial puncture within the past 1 week that does not easily compress the hemostatic site were included
8. ALT, AST, total bilirubin, direct bilirubin and indirect bilirubin exceeded the upper limit of normal value during screening visit
9. Positive test for human immunodeficiency virus (HIV-1 and HIV-2), hepatitis B surface antigen (HBsAg), anti-hepatitis C virus (anti-HCV) or syphilis at the Screening Visit.
10. Subjects who underwent surgery within 3 months before screening or schedule to have surgery during the trial, or those who have previously had surgery that may affect the PK profile or safety evaluation significantly of the study drug
11. Subjects who received any IMP within 3 months before the screening visit or planned to participate in other clinical trials during the trial
12. Received any drug that inhibits or induces liver metabolism of the drug within 1 month prior to screening visit
13. Received any prescription drugs (including vaccines) or non-prescription medications, and herbal supplements within 2 weeks prior to screening visit
14. Blood donation or blood loss≥200 mL within 3 month before screening, or schedule to donate blood during the trial or within 1 month after the end of the trial.
15. Had taken a special diet (including dragon fruit, mango, grapefruit, and/or xanthine diet, chocolate) and/or consumed excessive amounts of tea, coffee, grapefruit/grapefruit juice, and/or caffeinated beverages (averaging more than 8 cups per day of 200 ml each) in the 2 weeks prior to screening visit
16. History of alcohol abuse [more than 14 units of alcohol intake in one week (1 unit of alcohol equivalent to 285 mL of beer, 25 mL of spirits, or 100ml of wine), more than twice a week]
17. More than 10 cigarettes( or equivalent tobacco)per day in the 3 months prior to screening or unable to quit smoking during the trial period
18. Positive urine drug test at the Screening Visit History of drug abuse within the past 5 years
19. Pregnant or lactating women, or pregnancy test positive
20. Can not tolerate venipuncture or have a history of needle sickness and blood
21. Subjects with history of phlebitis
22. In the opinion of the Investigator, subjects should be excluded in this trial

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (AEs) | 8 +/- 1 days
Physical examination | 2 days
  Incidence of clinically significant physical examination findings
Vital signs | 2 days
  Incidence of clinically significant findings in systolic and diastolic blood pressure, heart rate and body temperature
12-lead electrocardiogram (ECG) | 24 hours
  Incidence of clinically significant findings in heart rate, PR interval, RR and QRS interval

IPD SHARING:
Plan to Share IPD: Undecided